CLINICAL TRIAL: NCT03393624
Title: Influence of Sleep Quality in Patients With Periorbicular Hyperchromia: a Case Control Study
Brief Title: Influence of Sleep Quality in Patients With Periorbicular Hyperchromia
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 150402
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Periorbital Disorder
Keywords: Dark circles; Periorbital hyperchromia; Sleep Quality; Facial aesthetics
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: patients with dark circles: Patients who believe they have periorbicular hyperchromia and have a confirmatory physical examination performed by a dermatologist.
- Controls: patients without dark circles: Patients who believe that they do not have periorbicular hyperchromia under their eyes and have physical examination that excludes dark circles carried out by a dermatologist.

SUMMARY:
Periorbital hyperchromia (POH) or periorbital hyperpigmentation, commonly known as "dark circles", is a relatively common condition and a frequent reason for dermatological consultation. It is defined as brown-colored pigmentation, ranging from light to dark, which mainly involves the lower eyelids. POH affects individuals over a wide age range, including both sexes and all ethnicities, and is associated with a tired and aged facial appearance. The most commonly affected people are those with the highest skin phototypes. Although the prevalence is similar between sexes and age groups, POH is a more frequent complaint in women. The dark circles characteristic of POH can negatively impact patients' quality of life, although it is not a condition associated with morbidity. Popularly it is believed that the poor quality of sleep is a factor responsible for its appearance, but there is no consistent data in the literature that prove this.

DETAILED DESCRIPTION:
We aim to compare the quality of sleep through the Pittsburgh Sleep Quality Index (PSQI-BR) already translated and validated in Portuguese for patients with periorbicular hyperchromia (cases) with patients without this complaint (controls) and to compare dermatological quality of life through the Quality of Life in Dermatology Index (DLQI) already translated and validated for Portuguese patients with periorbicular hyperchromia (cases) with patients without this complaint (controls). Patients and / or family members who consult in the Dermatology of the Hospital de Clínicas of Porto Alegre (preferably), but also other patients and / or relatives with outpatient care in this institution will be invited to participate in the control group.

The WinPepi program, version 11.32, was used to calculate the sample size. This objective predicts a Pareto Control Case study by age, with a ratio of 1: 1. The sample size was 252 subjects, 126 cases and 126 controls. Adding 10% to possible losses and refusals the sample size should be 280 subjects, with 140 cases and 140 controls. This value was stipulated taking into account the mean of 5.9 in the PSQI-BR of the cases already collected (n = 148 subjects) and corresponds to a difference of almost 3 points in the index ranging from zero to 21, corresponding to approximately 15% difference between groups. For this calculation was considered 80% power and significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Patients with periocular hyperchromia diagnosed by clinical examination.
* Controls: Patients without periocular hyperchromia diagnosed by clinical examination.

Exclusion Criteria:

* Pregnant patients
* Active collagenase patients
* Patients with bacterial or viral infections on the periorbicular area
* Patients undergoing any treatment modality for periocular hyperpigmentation in the last 3 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women over 18 years of age who agree to answer to quality of sleep and quality of life questionnaires. The "case" group should present periorbicular hyperchromia confirmed by physical examination and the group called "control" should not present periorbicular hyperchromia excluded by physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | at 1 day visit 1
  To evaluate the sleep quality in patients with periocular hyperpigmentation comparing with patients without periocular hyperpigmentation. The questionnaire consists of 19 questions, which are grouped into 7 components, with values distributed on a scale of zero to 3. These components are subjective quality of sleep, sleep latency, sleep duration, habitual sleep efficiency , sleep disorders, use of sleeping pills, and daytime dysfunction. The scores of these components are summed to form a global score, ranging from zero to 21. The higher the score, the worse the quality of sleep. A PSQI score> 5 indicates that the individual is experiencing major difficulties in at least 2 components, or moderate difficulties in more than 3 components.

SECONDARY OUTCOMES:
Quality of Life Index in Dermatology | at 1 day visit 1
  To evaluate the impact of periocular hyperpigmentation on patients' dermatological quality of life comparing with patients without periocular hyperpigmentation. this is a score used to evaluate the damage caused by dermatological diseases. It consists of 10 questions, with four alternative answers, corresponding to scores from 0 to 3. The maximum score is 30 and the minimum is zero, with 30 being the highest loss in the dermatological quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Boza, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rocha Barone C, Catucci Boza J, Challub Pires G, Perusato Pereira P, Ferreira Cestari T. The influence of sleep quality on the development of periocular hyperchromia: a case-control study. J Cosmet Dermatol. 2020 Jul;19(7):1760-1767. doi: 10.1111/jocd.13195. Epub 2019 Oct 30. PMID 31663247